CLINICAL TRIAL: NCT03301792
Title: Group Versus Traditional Prenatal Care for Diabetes: A Randomized Controlled Trial
Brief Title: Group Versus Traditional Prenatal Care for Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202209158
Record Dates: First submitted 2017-09-15; First posted 2017-10-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Gestational Diabetes; Type 2 Diabetes
Keywords: Group prenatal care; Diabetes
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Prenatal Care (No Intervention): Subjects randomized to routine care will receive their care in the usual diabetic clinic attended by residents and faculty. They will receive consultation with the diabetes educator at diagnosis and as needed. Patients are seen every 2 weeks (or more by provider discretion) until 37 weeks and weekly until delivery. Visits are 10-15 minutes and focus on routine screening tests and review of blood sugar logs/medication titration.
- Group prenatal care (Experimental): Group visits will be held every 2 weeks in a continuous cycle through a six session curriculum. Women will have weekly visits beginning at 37 weeks with traditional prenatal visits on the weeks when the group does not meet. Groups of 2-12 women will meet for two hour visits and much of that time will be spent on pregnancy, behavioral health, diabetes and nutrition education. Groups will be co-facilitated by a health educator and an obstetric provider. Women may be instructed to have additional visits in the traditional clinic at the discretion of the obstetric provider.
  Interventions: Behavioral: Group prenatal care

INTERVENTIONS:
Behavioral: Group prenatal care — Enrolled subjects will be randomly assigned in a 2:1 ratio to group or traditional care.
  Arms: Group prenatal care

SUMMARY:
The investigators primary objective is to conduct a randomized trial to determine the effect of diabetes group prenatal care on glycemic control and postpartum weight retention in women with type 2 diabetes and gestational diabetes.

DETAILED DESCRIPTION:
Long term, the investigator aims to test the central hypothesis that group prenatal care, compared to traditional prenatal care, will improve, 1.) glycemic control and, 2.) postpartum weight retention in women with type 2 and gestational diabetes. The objective of this proposal is to conduct a randomized trial in two phases to determine the effect of Diabetes Group Care (GC) on glycemic control in pregnant women with T2DM and GDM (Antepartum Phase) and the impact on postpartum weight retention (Postpartum Phase).

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. Type 2 diabetes OR gestational diabetes diagnosed by 2-step method(1) OR likely pre-existing Type 2 diabetes with one of the following during pregnancy and </= 34 weeks:

   1. 1 hour glucose challenge test >/= 185mg/dL OR
   2. A1c >/= 6.5% OR
   3. Fasting plasma glucose > 126mg/dL (2)
3. Ability to attend group prenatal visit at specified days and times
4. Willingness to be randomized at 22 weeks 0 days-34 weeks 0 days OR initial visit between 24 weeks 0 days-34 weeks 0 days
5. Ability to give informed consent

Exclusion Criteria:

1. Prior participation in diabetes group care
2. Type 1 Diabetes
3. Multiple gestation
4. Major fetal anomaly
5. Serious medical co-morbidity necessitating more care than can be safely provided in group setting, as deemed by medical provider.
6. Serious psychiatric illness including schizophrenia necessitating more care than can safely be provided in group setting, as deemed by medical provider.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Effect of Diabetes Group Care on maternal glycemic control | Initial study visit (22-34 weeks) through one year postpartum
  Determine the effect of Diabetes Group care on maternal glycemic control by randomizing women to Diabetes group care or traditional care and compare 1) Mean fasting blood glucose, 2) Mean 1-hour post-prandial blood glucose, and 3) Hemoglobin A1c at delivery, 4-12 weeks postpartum, six months postpartum, one year postpartum
Effect of Diabetes Group Care on postpartum weight retention | Pre-pregnancy weight (up to 6 months prior to initial visit) through one year postpartum
  Determine the impact of Diabetes Group care on postpartum weight retention in pounds based on postpartum weight retention at one year. Average weight retention will be compared at 4-12 weeks, six months postpartum, and one year postpartum.

SECONDARY OUTCOMES:
Completion of self-care activities | 37-39 weeks gestation
  Determine the effect of Diabetes Group care on maternal diabetes self-care activities by using the Diabetes Self-care Activities Scale (a measure of the number of days during the prior week in which the subject followed diet, exercise, blood sugar testing, and medication adherence recommendations)
Effect of Diabetes Group Care on number of blood glucose values | Initial study visit (22-34 weeks) through 39 weeks gestation
  Determine the effect of Diabetes Group care by measuring the percentage of recommended blood glucose values entered on logs since initial study visit
Maternal Antepartum Compliance | Initial study visit (22-34weeks) through 4-12 weeks postpartum
  Determine the effect of Diabetes Group Care on maternal antepartum compliance by assessing the number of prenatal appointments attended
Maternal Antepartum Physical Activity/Eating Behavior | Initial study visit (22-34weeks) through one year postpartum
  Determine the effect of Diabetes Group Care on maternal antepartum physical activity/eating behavior using a physical activity/eating behavior questionnaire
Maternal Antepartum Weight Gain | Initial study visit (22-34weeks) through delivery
  Determine the effect of Diabetes Group Care on maternal antepartum weight gain in pounds
Maternal Intrapartum Mode of Delivery | Delivery through 4-12 weeks postpartum
  Determine the effect of Diabetes Group Care on maternal intrapartum mode of delivery by assessing whether infant was delivered spontaneously, using vacuum, forceps, or cesarean.
Maternal Intrapartum Hypertensive Disease of Pregnancy | Delivery through 4-12 weeks postpartum
  Determine the effect of Diabetes Group Care on maternal intrapartum hypertensive disorders of pregnancy by assessing whether they develop gestational hypertension, preeclampsia, or eclampsia.
Maternal Postpartum Readmission | 4-12 weeks postpartum
  Determine the effect of Diabetes Group Care on maternal postpartum readmission by assessing number of maternal hospital readmissions within 6 weeks postpartum.
Maternal Postpartum Visit Attendance | 4-12 weeks postpartum
  Determine the effect of Diabetes Group Care on maternal postpartum visit attendance by assessing whether she attends a postpartum visit between 4-12 weeks postpartum.
Maternal Postpartum Glucose Testing | 4-12 weeks postpartum
  Determine the effect of Diabetes Group Care on maternal postpartum glucose testing
Maternal Postpartum Breastfeeding | 4-12 weeks postpartum, six months postpartum, one year postpartum
  Determine the effect of Diabetes Group Care on maternal postpartum breastfeeding using a breastfeeding scale questionnaire
Maternal Postpartum Contraception | 4-12 weeks postpartum, six months postpartum, one year postpartum
  Determine the effect of Diabetes Group Care on maternal postpartum contraception choices by assessing use of short acting reversible contraception, long acting reversible, and sterilization.
Neonatal Birthweight | delivery admission
  Determine the effect of Diabetes Group Care on neonatal birth weight in grams
Neonatal Gestational Age | delivery admission
  Determine the effect of Diabetes Group Care on neonatal gestational age at delivery
Neonatal APGAR Scores | delivery admission
  Determine the effect of Diabetes Group Care on neonatal APGAR score
Neonatal Adiposity and body composition | delivery admission through one year postpartum
  Determine the effect of Diabetes Group Care on neonatal adiposity and body composition by air displacement plethysmography within 1 week of delivery. Skin fold thickness of triceps, subscapular, ilium, and thigh at delivery, six weeks, six months, one year postpartum.
Neonatal body measurements-Weight | delivery through one year postpartum
  Determine the effect of Diabetes Group Care on neonatal weight in grams
Neonatal body measurements-Length | delivery through one year postpartum
  Determine the effect of Diabetes Group Care on neonatal length in centimeters
Neonatal body measurements-Head Circumference | delivery through one year postpartum
  Determine the effect of Diabetes Group Care on neonatal head circumference in centimeters
Neonatal NICU Admission | delivery admission
  Determine the effect of Diabetes Group Care on neonatal NICU admission
Neonatal Hypoglycemia | delivery admission
  Determine the effect of Diabetes Group Care on neonatal hypoglycemia
Neonatal Outcomes | delivery admission
  Determine the effect of Diabetes Group Care on neonatal hematocrit
Neonatal Jaundice | delivery admission
  Determine the effect of Diabetes Group Care on neonatal jaundice
Neonatal Stillbirth Rates | delivery admission
  Determine the effect of Diabetes Group Care on neonatal stillbirth rates
Psychosocial Stress | Initial study visit (22-34weeks) through one year postpartum
  Determine the effect of Diabetes Group Care on psychosocial stress by comparing Cohen's Perceived Stress at study entry visit, last study visit (37-39 weeks) and 4-12 weeks postpartum, six months postpartum, one year postpartum.
Psychosocial Stress | Initial study visit (22-34weeks) and six months postpartum
  Determine the effect of Diabetes Group Care on psychosocial stress by comparing life events checklist at study entry visit and six months postpartum
Psychosocial Distress | Initial study visit (22-34 weeks) through 4-12 weeks postpartum
  Determine the effects of Diabetes Group Care on psychosocial stress by comparing Pregnancy Distress questionnaire at study entry, last study visit (37-39 weeks), and 4-12 weeks postpartum
Psychosocial Anxiety | Initial study visit (22-34weeks) through one year postpartum
  Determine the effects of Diabetes Group Care on psychosocial stress by comparing GAD-7 at study entry, last study visit (37-39weeks) and 4-12 weeks postpartum, six months postpartum, one year postpartum.
Psychosocial Depression | Initial study visit (22-34weeks) through 1 year postpartum
  Determine the effects of Diabetes Group Care on depression by comparing the Edinburgh Postnatal Depression Scale at study entry, last study visit (37-39 weeks) and 4-12 weeks postpartum, six months postpartum, one year postpartum
Psychosocial Stress and Depression | Delivery through postpartum
  Determine the effects of Diabetes Group Care on stress and depression by measuring alcohol or drug use in first year postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Megan Lawlor, MD, Principal Investigator — Assistant Professor, Washington University in St. Louis
Locations (2):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - University of Utah, Salt Lake City, Utah